CLINICAL TRIAL: NCT03537157
Title: A Phase II, Multicentre, Double-blind, Randomised, Placebo-controlled Study of Rifaximin Delayed Release 400 mg Tablet: Clinical Efficacy and Safety in the Prevention of Post-operative Endoscopic Crohn's Disease Recurrence
Brief Title: A Multicentre Study on Rifaximin in Post-operative Endoscopic Crohn's Disease Recurrence Prevention
Acronym: STOP-PER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The decision to prematurely close the trial recruitment period was taken due to the difficulties in the recruitment of patients. This decision has not been triggered by any unexpected safety signals identified during the study conduction.
Sponsor: Alfasigma S.p.A. (Industry)
Collaborators: Cromsource (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RETIPC/01/17
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-07

CONDITIONS: Crohn Disease
Keywords: Crohn Disease recurrence
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: The study is a multicentre, randomised, double-blind, placebo controlled trial to assess the efficacy and safety of Rifaximin delayed release 400 mg tablet (800 mg BID daily) administered for 26 weeks in the prevention of endoscopic Crohn's disease recurrence following ileocolonic resection, in patients who had undergone curative ileocolonic resection, with ileocolonic anastomosis for Crohn's disease.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active drug will be masked with a placebo identical to the active drug. Patients will be identified by a code and central readers will not have access to the administered treatments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifaximin delayed release tablets (Experimental): Two 400 mg tablets twice a day (total daily dose 1600 mg) for 26 weeks
  Interventions: Drug: Rifaximin delayed release tablets
- Placebo (Placebo Comparator): Two placebo tablets twice a day for 26 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rifaximin delayed release tablets — Active intervention
  Arms: Rifaximin delayed release tablets
Other: Placebo — Comparator placebo
  Arms: Placebo

SUMMARY:
Crohn's Disease (CD) is a chronic pathology characterized by exacerbations and remissions. Recurrent inflammation can cause bowel strictures, fistulae (often perianal) or abscesses. CD often requires intestinal resection. Surgery in CD is not curative, Therefore, endoscopic follow-up 6-12 months after surgery is recommended. Given the association between enteric bacteria and postoperative CD recurrence, antibacterial agents were shown to be effective in reducing the severity of endoscopic recurrence, but prolonged administration causes significant toxicity. The efficacy of "systemic antibiotics" and the experimental evidence of the central role of luminal flora as an essential factor in the development of post chirurgic CD recurrence provide the rationale for evaluating a locally acting antibiotic like Rifaximin.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic, relapsing, remitting, systemic disease, which may result in transmural inflammation of the gastrointestinal tract. The precise aetiology is unknown: it is a lifelong disease arising from an interaction between genetic and environmental factors, but predominantly observed in developed countries of the world. CD can affect the entire digestive tract from the mouth to the anus, but the most commonly affected sites are the ileum and the ascending colon . The clinical course of CD is characterized by exacerbations and remissions. Therefore, recurrent inflammation can cause bowel strictures, fistulae (often perianal) or abscesses. Moreover, Crohn's disease (CD) often requires intestinal resection, despite treatment with immunosuppressive and biologic therapies.

Surgery in CD is not curative, and post-operative recurrence (POR) is a frequent event. Historically, up to 70% of patients who undergo CD-related resection develop postoperative endoscopic recurrence at or proximal to the surgical anastomosis within 1 year and approximately one-third of patients with CD, who have a first resection, require a second within 10 years.

Endoscopic lesions usually precede and correlate with future clinical recurrence (about 20-25% per year), and predict the development of Crohn's disease-related complications and the need for re-intervention.

Therefore, endoscopic follow-up 6-12 months after surgery is recommended. Given the association between enteric bacteria and postoperative CD recurrence, antibacterial agents directed against anaerobic bacteria (ornidazole and metronidazole) were shown to be effective in reducing the severity of endoscopic recurrence, but prolonged administration (more than 3 months) of these antibiotics causes significant toxicity, mainly neuropathy and gastrointestinal intolerance. The efficacy of "systemic antibiotics" and the experimental evidence of the central role of luminal flora as an essential factor in the development of post chirurgic CD recurrence provide the rationale for evaluating a locally acting antibiotic like Rifaximin in this condition.

ELIGIBILITY:
Inclusion Criteria:

* Crohn Disease with curative ileocolonic resection
* Randomization within 45 days from ileocolonic resection or end or loop ileostomy within last year and closure occurred within 45 days from randomization
* Fecal stream restoration at least 14 days prior to randomization
* Presence of at least one risk factor for recurrence
* Pregnancy protection on board during the study for childbearing female subjects

Exclusion Criteria:

* Presence of CD proximally or distally to the site of resection
* Patients with strictureplasties at index surgery or ileorectal anastomosis
* patients with active perianal CD
* Patient treated with other treatments usually utilised for CD
* Patients with active diseases with gastrointestinal involvement
* intestinal obstruction or pseudo-obstruction
* Patients presenting diarrhoea plus fever or bloody stools
* Positivity to clostridium difficile toxin
* Severe hepatic or renal impairment
* Presence of severe cardiac insufficiency
* Hypersensitivity to rifamycin antimicrobial agents
* other conditions that would interfere or prevent the study completion
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
Rutgeerts score | 26 weeks
  Rate of patients presenting a rutgeerts score higher than or equal to i2 will be considered as endpoint. Endoscopic remission will be defined as a Rutgeerts score of i0 or i1 and recurrence defined as a Rutgeerts score of ≥i2 (i0, no lesions; i1, ≤5 aphthous lesions; i2, >5 aphthous lesions or anastomotic ulcer <1 cm; i3, diffuse aphthous ileitis with diffusely inflamed mucosa; i4, diffuse inflammation with large ulcers, nodules, and/or narrowing) at the anastomosis and neoterminal ileum. (Rutgeerts P, 1990)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grimaldi, MD, Study Director — Alfasigma S.p.A.
Locations (1):
- Humanitas Clinical Research Center, Rozzano, Italy

IPD SHARING:
Plan to Share IPD: No